CLINICAL TRIAL: NCT00673933
Title: A Blinded, Randomized, Intra-individual, Vehicle-controlled and Multi-centre Study of Photodynamic Therapy With MAL Cream in Patients With Skin Type V or VI With Acne Vulgaris
Brief Title: Photodynamic Therapy (PDT) With Methyl Aminolevulinate (MAL) Cream in Patients With Skin Type V or IV With Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Photocure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PC TA203/08
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2013-07-12 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — methyl 5-aminolevulinate; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): PDT using MAL crem
  Interventions: Drug: Methyl aminolevulinate (MAL) PDT
- 2 (Placebo Comparator): PDT using Placebo cream
  Interventions: Drug: Methyl aminolevulinate (MAL) PDT

INTERVENTIONS:
Drug: Methyl aminolevulinate (MAL) PDT — Cream application followed by illumination with red light

SUMMARY:
In this multicenter study, patients with dark skin and acne vulgaris will be included. The patients will receive treatment with MAL PDT and placebo PDT.

DETAILED DESCRIPTION:
The treatment period started within 2 weeks of the study screen. Patients received two treatments (MAL PDT and vehicle PDT) to each of the treatment areas, 2 weeks apart, and were followed-up 4 weeks after last treatment. The total duration of the study was 6-8 weeks.

Methyl aminolevulinate 80 mg/g cream (MAL cream 8%)and vehicle was applied for 1.5 hours before illumination (Aktilite® CL128), total light dose 37 J/cm2

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients, age 15 to 40 years with acne vulgaris.
2. Patients with skin type V or VI (Fitzpatrick).
3. Patients with two areas of each 8x8 cm2 on the back that include at least 5 inflammatory lesions (papules, pustules, and nodules) each. The minimum distance between the two areas should be at least 4 cm.
4. Patients with no more than 2 nodular lesions in any of the two areas of each 8x8 cm2 on the back.
5. Patients who are surgically sterile, postmenopausal, abstinent, or willing to use an adequate means of contraception including birth control pills, or barrier methods and spermicide for at least 14 days prior to Day 0. Patients using birth control pills must have used the same product and dose for at least 3 months and must agree to stay with the same product and dose for an additional 3 months.
6. Patients must be willing and capable of following study instructions to the extent and degree required by the protocol.
7. Patients must sign the approved informed consent form prior to any study procedures.
8. Patients must be willing to be photographed. Patients must be willing to sign a photography consent form.

Exclusion Criteria:

1. Known allergy to MAL, to a similar PDT compound, or to excipients of the cream.
2. Participation in other clinical studies either concurrently or within the last 30 days.
3. Patients who have a condition or who are in a situation, which, in the investigator's opinion, may put the patient at risk, may confound the study results, or may interfere with the patient's participation in the study.
4. Clinically significant sensitivity to visible light, or has porphyria or porphyrin sensitivity.
5. Exposure to ultraviolet radiation (UVB phototherapy) within the last 30 days.
6. Patients with a washout period for topical treatments for their acne in the two treatment areas of less than 14 days. Any topical treatment on the face or other areas outside the two treatment areas will be allowed.
7. Patients with a washout period for oral antibiotics for treatment of their acne of less than 1 month.
8. Patients with a washout period for oral isotretinoin of less than 6 months.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2008-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashish C Bhatia, MD, Principal Investigator — Dermatology Institute of DuPage Medical Group
Locations (2):
- United States (2):
  - DuPage Medical Group, Naperville, Illinois
  - Academic Dermatology Associates, Albuquerque, New Mexico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two areas on the back per patient was treated, one area with Visonac and one with vehicle
Groups:
- Visonac Cream With PDT and Vehicle and PDT: Two areas on the back per patient was treated, one area with Visonac and one with vehicle. Methyl aminolevulinate (MAL) PDT : Cream application followed by illumination with red light
Period: Overall Study
Arm/Group | Visonac Cream With PDT and Vehicle and PDT
Started | 20
Completed | 17
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Visonac and Vehicle Cream With PDT: Two areas on the back per patient was treated, one area with Visonac (Methyl aminolevulinate) and one with vehicle followed by red light illumination.
Arm/Group | Visonac and Vehicle Cream With PDT
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 16
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 20
Skin type [Number; unit: participants] — Skin type according to the Fitzpatrick Classification Scale. Skin type V: Brown, dark brown.Very rarely burns, tans very easily Skin type VI: Black, very dark brown to black. Never burns, tans very easily, deeply pigmented
  participants
    Skin type V | 18
    Skin type VI | 2
Inflammatory lesions [Mean (Full Range); unit: lesion]
  Visonac treated area | 5.9 [5 to 11]
  vehicle treated area | 6.0 [5 to 10]
Non inflammatory lesions [Mean (Full Range); unit: Lesion]
  Visonac treated area | 6.5 [1 to 21]
  vehicle treated area | 5.4 [2 to 17]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Moderate to Severe Hypopigmentation and Hyperpigmentation Assessed After Treatment
Time Frame: 4 weeks after last treatment, 6 weeks after baseline
Measure: Number; unit: participants
Groups:
- Visonac Cream With PDT: PDT using MAL cream
  Methyl aminolevulinate (MAL) PDT : Cream application followed by illumination with red light
- Vehicle Cream With PDT: PDT using Placebo cream
  Methyl aminolevulinate (MAL) PDT : Cream application followed by illumination with red light
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 20 | 20
participants | 0 | 0

2. Secondary Outcome: Erythema Score (Mild and Moderate)Immediately After First PDT
Description: Patients with mild or moderate erythema after first treatment at baseline.
Time Frame: Immediately after treatment at baseline
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 20 | 20
percentage of participants | 10.5 | 0.0

3. Secondary Outcome: Change in Inflammatory Lesion Counts From Baseline
Time Frame: 4 weeks after last treatment, 6 weeks after baseline
Population: ITT
Measure: Mean (Standard Deviation); unit: lesion count
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 20 | 20
lesion count | -3.70 (2.43) | -3.90 (2.07)

4. Secondary Outcome: Change in Noninflammatory Lesion Counts From Baseline
Time Frame: 4 weeks after last treatment, 6 weeks after baseline
Population: ITT
Measure: Mean (Standard Deviation); unit: lesion count
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 20 | 20
lesion count | -2.95 (4.84) | -2.50 (2.65)

5. Secondary Outcome: Erythema Score (Mild and Moderate)Immediately After Second Treatment
Description: Patients with mild or moderate erythema after second treatment.
Time Frame: Immediately after second treatment, 2 weeks after baseline
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 20 | 20
percentage of participants | 11.1 | 0

6. Secondary Outcome: Erythema Score (Mild and Moderate)1 Day After First Treatment
Description: Patients with mild or moderate erythema 1 day after first treatment.
Time Frame: 1 day after 1st treatment and baseline
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Number analyzed (Participants) | 20 | 20
percentage of participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Visonac Cream With PDT | Vehicle Cream With PDT
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 12/20 | 12/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Visonac Cream With PDT (N=20) | Vehicle Cream With PDT (N=20)
Paraesthesia (Nervous system disorders) | 1 (1) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pruritus nos (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Skin warm (Skin and subcutaneous tissue disorders) | 7 (9) | 5 (5)
Hematoma Nos (Vascular disorders) | 1 (1) | 1 (1) — Non treatment site, included under both Visonac and vehicle arm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days